CLINICAL TRIAL: NCT03781622
Title: WOLF - Prospective Feasibility Clinical Investigation to Evaluate the Safety and Technical Performance of the WOLF Thrombectomy Device in Acute Ischemic Stroke Patients
Brief Title: WOLF - Feasibility Neurothrombectomy Study in Acute Ischemic Stroke Patients
Acronym: WOLF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: 880 Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 0001-CAN
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, multi-center, feasibility clinical investigation to evaluate the safety and device technical performance of the WOLF Thrombectomy Device in removing thrombus from an occluded large intracranial vessel(s) in patients with acute ischemic stroke. The device may be used alone or as an adjunct to intravenous tissue plasminogen activator (tPA) and/or to other traditional, thrombectomy modalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- WOLF Thrombectomy Device Arm (Experimental): Patients enrolled in the study who received the treatment and who met all Inclusion and Exclusion Criteria
  Interventions: Device: WOLF Thrombectomy Device

INTERVENTIONS:
Device: WOLF Thrombectomy Device — Mechanical thrombectomy for the neurovasculature

SUMMARY:
This study is being conducted as a feasibility clinical investigation to collect safety and technical performance data of the WOLF Thrombectomy Device for the removal of thrombus in the neurovasculature.

DETAILED DESCRIPTION:
This study has been designed as a prospective, non-randomized, multi-center, feasibility clinical investigation to evaluate the safety and device technical performance of the WOLF Thrombectomy Device in removing thrombus from an occluded large intracranial vessel(s) in patients with acute ischemic stroke. The device may be used alone or as an adjunct to intravenous tissue plasminogen activator (tPA) and/or to other traditional, thrombectomy modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥18 years (no upper limit).
2. NIHSS > 6 at the time of baseline neuro imaging.
3. Endovascular treatment intended to be initiated within 60 minutes of qualifying neuroimaging and intended vessel recanalization within 90 minutes of qualifying neuroimaging.
4. Stroke symptom onset within 24hrs of when groin puncture can be obtained.
5. Anterior and posterior circulation large vessel occlusion as confirmed through neuro imaging (CT/CTA/mCTA/MRI/MRA).
6. Neurovascular imaging (CTA/mCTA and or MRA) must include the aortic arch, cervical vessels and intracranial circulation.
7. Advanced neurovascular imaging is required for patients when groin puncture can be obtained after 6 hours and before 24 hours (multiphase CTA, CT Perfusion or perfusion diffusion imaging).
8. The occlusion is located in a proximal intracranial artery (carotid artery, M1 segment of the MCA, or proximal M2 divisions) of the anterior circulation for patients after 6 hours and before 24 hours.
9. There is imaging and clinical evidence of small core and large areas at risk, defined in the previous trials (DAWN & DEFUSE 3) as either:

   i. NIHSS ≥10 and either 0-21 ml core infarct (≥80 years old) or 0-31 ml core infarct (<80 years old), or NIHSS≥20 and 31 to <51ml core infarct and <80 years old (DAWN trial criteria).

   OR ii. Ischemic core volume is < 70 ml, mismatch ratio is >/= 1.8 and mismatch volume* is >/= 15 ml (DEFUSE 3 trial criteria).
10. Pre-stroke disability limited to patients with mRS ≤ 2.
11. Written informed consent to participate given by subject or legal / authorized representative per local ethics committee requirements.

Exclusion Criteria:

1. Female subject is known to be pregnant.
2. Absence of large vessel occlusion on neuro imaging.
3. Presence of existing or preexisting large vessel infarction.
4. Angiographic evidence of excessive arterial tortuosity or access that precludes the WOLF device from reaching the thrombus.
5. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR >2.5.
6. Patient has a known hypersensitivity to contrast media.
7. Medical reasons the procedure cannot be performed (i.e. patient is experiencing active, uncontrolled bleeding, etc.)
8. Subject is known to be currently enrolled in another investigational trial that could interfere with the endpoint analysis of this trial.
9. ASPECT < 5 or > 1/3 MCA vascular territory compromised as evidenced by CT or MRI.
10. Significant mass effect and mid-line shift.
11. Any evidence of intracranial hemorrhage on imaging.
12. For posterior circulation large vessel occlusion evidence of completed significant brain stem infarction.
13. Posterior circulation after 6 hours.
14. Patients are known to have severe psychiatric disorders, substance abuse, or other reason for being unable to follow trial follow-up instructions.
15. Subject has a known significant concomitant illness with a life expectancy of <6 months.
16. Subject has a known allergy to nickel.
17. Subject has a known history of severe intracranial atherosclerotic disease (ICAD).
18. Subject is unlikely to be able and willing to comply with site standard medical follow up to 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Primary Technical Success Endpoint | At index procedure
  Technical Success defined as the ability to achieve a revascularization rate (Thrombolysis in cerebral infarction [TICI] 2b/3) of ≥50% with the first pass of the WOLF Thrombectomy device. Revascularization is assessed by the investigator using fluoroscopy and after the first pass of the device is assessed using the TICI scale. Additional passes will be performed as necessary and the total number of attempts to achieve revascularization documented.
Primary Safety Endpoint | At index procedure and through 24 hours post procedure.
  WOLF device-related adverse events (incidence, relationship to device and severity) at index procedure and through 24 hours post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Brian van Adel, MD, Principal Investigator — Hamilton General Hospital
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No